CLINICAL TRIAL: NCT05549362
Title: Dietary Approaches to Longevity and Health
Brief Title: DiAL Health Research Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2021-020
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Aging; Weight Loss; Treatment Adherence
MeSH Terms: conditions — Weight Loss; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ad libitum Control (Placebo Comparator): No treatment control condition.
  Interventions: Other: Dial Health Research Study
- Traditional CR (Active Comparator): A 25% calorie restriction (CR) intervention delivered via traditional in-person sessions.
  Interventions: Other: Dial Health Research Study
- Adaptive CR (Active Comparator): A 25% calorie restriction (CR) intervention delivered via a remote, adaptive, and technology-driven intervention program.
  Interventions: Other: Dial Health Research Study
- Traditional TRE (Active Comparator): An eight-hour time restricted eating (TRE) intervention delivered via traditional in-person sessions.
  Interventions: Other: Dial Health Research Study
- Adaptive TRE (Active Comparator): An eight-hour time restricted eating (TRE) intervention delivered via a remote, adaptive, and technology driven intervention program.
  Interventions: Other: Dial Health Research Study

INTERVENTIONS:
Other: Dial Health Research Study — To evaluate the feasibility and efficacy of dietary intervention approaches to slow mechanisms of aging.

SUMMARY:
The purpose of this study is to conduct a five-arm pilot and feasibility trial in healthy, young individuals without obesity to evaluate the feasibility and efficacy of dietary intervention approaches to slow mechanisms of aging.

DETAILED DESCRIPTION:
Nutritional interventions are one of the most promising non-pharmacological approaches that attenuate aging. Continuous calorie restriction (CR), the most studied intervention, extends lifespan in animals and, in humans, slows biological aging and improves healthspan (e.g., disease risk factors, quality of life). In the largest clinical trial of CR in humans (CALERIE 2), adherence to 25% CR waned to ~12% CR over 2 years, which questions the practicality of such interventions over longer periods. CALERIE 2, however, did not benefit from a more advanced approach, namely a Just-in-Time Adaptive Intervention (JITAI), which tailors and optimizes the intervention for each subject. JITAIs strive to provide individuals with the right type and amount of personalized support when necessary by adapting the intervention delivery to the present adherence, needs and environment of the subject. This is accomplished by the use of mobile health (mHealth) technology (smartphones, sensors) to objectively evaluate intervention adherence in real-time and to adapt intervention delivery to each individual over time. The near real-time collection of ecologically valid and objective data from people in their free-living environment dramatically improves the ability to promote adherence and subject engagement.

Newer approaches, such as time-restricted eating (TRE), where food intake is restricted to less than a 10-hour period of the day, may also benefit aging. Short-term pilot studies of TRE showed that, independent of CR, eating over a 6-hour window that began in the morning significantly improved diabetes and cardiovascular risk factors (healthspan) and biomarkers of primary aging (e.g., autophagy, oxidative stress, nutrient sensing). The long-term feasibility of TRE is unknown, and it is unclear if TRE interventions with JITAI designs enhance intervention feasibility and adherence in the context of healthy aging.

The current trial will examine the feasibility and preliminary efficacy of two CR and two TRE interventions to modulate healthspan and biomarkers of aging in healthy, young (25-45 years) individuals. In a 5-arm pilot and feasibility trial, 90 people without obesity (BMI 22-29.9 kg/m2) will be randomized to either ad libitum Control, Traditional CR, Adaptive CR, Traditional TRE, or Adaptive TRE for 24 weeks (n=18/group) for six months

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant pre-menopausal female, 25-45 years of age, inclusive
2. BMI ≥22kg/m2 and <30kg/m2
3. Screening lab values within normal limits, or deemed not clinically significant
4. Stable body weight (less than ± 2kg) in the past 6 months
5. Regularly wake up between 5-8 AM

Exclusion Criteria

1. History of prior bariatric surgery, active gallstone disease, extensive bowel resection or any disease or condition that seriously affects body weight and/or body composition
2. Regular (daily) use of medications for chronic medical conditions.
3. History or clinical manifestation of:

   1. Significant chronic metabolic, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, immune, hepatic, renal, urologic, circadian, sleep disorders, reproduction or other condition that would not be considered 'healthy' in opinion of the investigator
   2. Anemia (Hb <10 g/dL or hematocrit < 30)
   3. Diabetes or fasting glucose ≥ 126 mg/dL or HbA1c ≥ 6.5% at screening
   4. Hypertension (Systolic Blood Pressure >140 mmHg & Diastolic Blood Pressure >90 mmHg)
   5. Cancer requiring treatment in the past 5 years (except for non-melanoma skin cancer)
   6. Low Bone mineral density z-score < -2.0 of the hip (total hip or femoral neck) or lumbar spine (L1-L4)
   7. Depression as determined by the Beck Depression Inventory-II > 19
   8. Pregnant, postpartum (< 12 months) or lactating females or attempting to become pregnant in the next 7 months
   9. Current or history (within the past 5 years) of an eating disorder
   10. Asthma or sleep apnea
4. Lifestyle related factors that would confound outcomes:

   1. Non-conventional eating patterns (vegan, paleo, fasting, etc.) and eating duration (<11 hours per day)
   2. Drug or alcohol abuse (up to 14 drinks a week are allowed) within the past 2 years
   3. Current smoking, vaping or use of tobacco products within the past 6 months
   4. Currently participating or recently engaged (4 consecutive weeks in the past 3 months) in heavy aerobic activity (e.g., jogging, running, or riding fast on a bicycle) ≥ 240 minutes per week or heavy resistance training ≥ 3 times per week that results in heavy breathing and sweating.
   5. Perform overnight shift work > 1 day/week or plan to cross more than 2 time zones within 1 month of study assessments
5. Unwilling or unable to adhere to the rigors of the protocol or failure to complete the behavioral run-in task (at least 80% compliance)

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intervention satisfaction ratings | 6 months
  Intervention satisfaction will be assessed via Likert ratings for each study group.
Percent CR (CR groups only) | 6 months
  Percent calorie restriction (CR) will be quantified for the 2 CR groups via doubly labeled water and the intake balance method.
Percent adherence to TRE (TRE groups only) | 10 days over at least 3 timepoints
  Percent adherence to the eating window in the time-restricted eating groups will be assessed by continuous glucose monitoring.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana

IPD SHARING:
Plan to Share IPD: Yes
Researchers are encouraged to contact the PIs to request study data.
Supporting Information: Study Protocol
Time Frame: Following data collection, data cleaning, data lock, data analysis, and submission of the primary outcome paper.
Access Criteria: An institutional signing official from the researcher's institution is required to execute a Data Transfer Agreement.